CLINICAL TRIAL: NCT04040686
Title: Technetium-99m Labeled Anti-HER2 sdAb (99m-Tc-NM-02) for HER2 Expression Detection in Breast Cancer
Brief Title: HER2 Expression Detection in Breast Cancer Using 99mTc-NM-02
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: NanoMab Technology (UK) Limited (Industry)
Responsible Party: Principal Investigator, Zhao Jin Hua, MD, Director Department of Nuclear Medicine, Principal Investigator, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [2019]52
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: HER2; single domain antibody (sdAb); SPECT/CT imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of 99mTc-NM-02 (Experimental): All breast cancer patients recruited to the study will be administered 3-12 MBq/kg of 99m-Tc-NM-02 (99m-Tc labeled anti-HER2 sdAb) in a single dose injection
  Interventions: Drug: Injection of 99mTc-NM-02

INTERVENTIONS:
Drug: Injection of 99mTc-NM-02 — Patient will be injected with microdose (<100ug) of 99mTc-NM-02 radiotracer
  Other Names: anti-HER2 SPECT/CT radiotracer

SUMMARY:
A 99mTc-labeled anti-HER2-sdAb (99mTc-NM-02) will be developed for SPECT/CT assessment of HER2 expression in breast cancer patients. Its safety, radiation dosimetry and biodistribution, and the relationship between tumor uptake and HER2 immunohistochemistry results will be investigated.

DETAILED DESCRIPTION:
To evaluate the safety, dosimetry and efficacy of 99m-Tc labeled anti-HER2 single domain antibody (sdAb) (Product Code Name: 99mTc-NM-02) SPECT/ CT imaging of HER2 expression in Breast Cancer and compare it with the existing gold standard " HER2 expression detection" by biopsy tissue immunohistochemistry (IHC) and/or Fluorescence In Situ Hybridization (FISH) method. It is also to establish a new clinical method of non-invasive HER2 expression detection in breast cancer using 99m-Tc labeled anti-HER2 sdAb

ELIGIBILITY:
Inclusion Criteria:

1. Adult female, age 18 years or older
2. Prior diagnosis of breast cancer
3. Willing to participate in this study and given written informed consent
4. AST, ALT, BUN, Cr not more than double the normal values
5. Subjects of childbearing potential must be willing to undergo a pregnancy test prior to enrolment

Exclusion Criteria:

1. Pregnancy (subjects with a positive pregnancy test at baseline screening period or who are planning to become pregnant during the study period)
2. Breastfeeding (subjects in lactation)
3. No biopsy tissue sample can be provided for HER2 expression detection
4. Subjects with pacemakers
5. Hepatitis B virus infection (including carriers) at screening, ie hepatitis B surface antigen (HBsAg) positive, or hepatitis C antibody (anti-HCV) positive, or acquired immunodeficiency disease (HIV) infected, or serum syphilis positive person
6. Abnormal liver function during baseline screening period : AST or ALT> 2 times the upper limit of normal value (ULN), if the marginal increase of a single index is judged as having no clinical significance by the investigator, it can be retested during the screening period. Once, if ≤ 2 times ULN after retesting, consider enrolling).
7. Impaired renal function during screening: serum creatinine or urea nitrogen > 1.5 times ULN.
8. Within 4 months prior to the baseline screening period , myocardial infarction or other cardiac events requiring hospitalization (unstable angina, etc.), cerebrovascular accident, transient ischemic attack, acute congestive Heart failure or severe arrhythmia (ventricular arrhythmia, atrioventricular block above II)
9. Subjects with pulmonary embolism or deep vein thrombosis
10. Various infections that the investigators consider unsuitable for study, including but not limited to patients with various infections requiring further treatment, such as urinary tract infections, respiratory infections, and diabetic foot infections.
11. Patients with abnormal thyroid function during baseline screening period (including but not limited to active hyperthyroidism, hypothyroidism or Hashimoto's thyroiditis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Assessment of HER2 expression in Breast cancer using 99mTc-NM-02 SPECT/CT Scan | 1 year
  Visual analysis will be carried out by 4 experienced nuclear medicine physicians to observe the uptake of 99m-Tc-NM-02 in breast malignant lesions. A 4 point system will be used to interpret the scans for abnormalities. It is categorised as such: score 0, no abnormal increased uptake; score 1, low increased uptake; score 2, moderate increased uptake; score 3, high increased uptake. The lesion will be considered positive for malignancy if the score is 2 or higher.
Semiquantitative Assessment of Breast and other Metastatic Lesions in 99mTc-NM-02 SPECT/CT Scan | 1 year
  Each subject will be administered 3-12 MBq/kg of 99mTc-NM-02 and the semiquantitative analysis of the region of interest (ROI) will be performed in breast and other metastatic lesions. Higher level of HER2 expression (Tumor proportion score, TPS), higher ROI in tumor.
Safety of 99mTc-NM02 through Adverse Event Monitoring | 2 days
  Subjects will be observed for safety after administration of 99mTc-NM-02, and will do follow up at 48h p.i. Subjects will do blood test to observe for abnormalities in clinical parameters and compare to baseline results.
Safety of 99m-Tc-NM-02 through Adverse Event Monitoring | 7 days
  Subjects will be observed for safety after administration of 99mTc-NM-02, and will do follow up at 7d p.i. Subjects will be contacted by investigator by phone and asked several questions related to subject's health after 99m-Tc-NM-02 injection and concomitant drugs.

SECONDARY OUTCOMES:
HER2 Expression Heterogeneity | 1 year
  Biopsy tissue sample IHC and FISH HER2 test results from subject's primary tumor will indicate its HER2 expression level, this results will be compared with our radiotracer uptake in the primary tumor and will look for heterogeneity while observing for uptake in other metastatic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Zhao, PhD, Principal Investigator — Shanghai General Hospital Nuclear Medicine Dept
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Ni J, Ramkissoon SH, Xie S, Goel S, Stover DG, Guo H, Luu V, Marco E, Ramkissoon LA, Kang YJ, Hayashi M, Nguyen QD, Ligon AH, Du R, Claus EB, Alexander BM, Yuan GC, Wang ZC, Iglehart JD, Krop IE, Roberts TM, Winer EP, Lin NU, Ligon KL, Zhao JJ. Combination inhibition of PI3K and mTORC1 yields durable remissions in mice bearing orthotopic patient-derived xenografts of HER2-positive breast cancer brain metastases. Nat Med. 2016 Jul;22(7):723-6. doi: 10.1038/nm.4120. Epub 2016 Jun 6. PMID 27270588
- [Background] Burstein HJ. The distinctive nature of HER2-positive breast cancers. N Engl J Med. 2005 Oct 20;353(16):1652-4. doi: 10.1056/NEJMp058197. No abstract available. PMID 16236735
- [Background] Arteaga CL, Sliwkowski MX, Osborne CK, Perez EA, Puglisi F, Gianni L. Treatment of HER2-positive breast cancer: current status and future perspectives. Nat Rev Clin Oncol. 2011 Nov 29;9(1):16-32. doi: 10.1038/nrclinonc.2011.177. PMID 22124364
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Background] Gingras I, Gebhart G, de Azambuja E, Piccart-Gebhart M. HER2-positive breast cancer is lost in translation: time for patient-centered research. Nat Rev Clin Oncol. 2017 Nov;14(11):669-681. doi: 10.1038/nrclinonc.2017.96. Epub 2017 Aug 1. PMID 28762384
- [Background] Loibl S, Gianni L. HER2-positive breast cancer. Lancet. 2017 Jun 17;389(10087):2415-2429. doi: 10.1016/S0140-6736(16)32417-5. Epub 2016 Dec 7. PMID 27939064
- [Background] Niikura N, Liu J, Hayashi N, Mittendorf EA, Gong Y, Palla SL, Tokuda Y, Gonzalez-Angulo AM, Hortobagyi GN, Ueno NT. Loss of human epidermal growth factor receptor 2 (HER2) expression in metastatic sites of HER2-overexpressing primary breast tumors. J Clin Oncol. 2012 Feb 20;30(6):593-9. doi: 10.1200/JCO.2010.33.8889. Epub 2011 Nov 28. PMID 22124109
- [Background] Baum RP, Prasad V, Muller D, Schuchardt C, Orlova A, Wennborg A, Tolmachev V, Feldwisch J. Molecular imaging of HER2-expressing malignant tumors in breast cancer patients using synthetic 111In- or 68Ga-labeled affibody molecules. J Nucl Med. 2010 Jun;51(6):892-7. doi: 10.2967/jnumed.109.073239. Epub 2010 May 19. PMID 20484419
- [Background] D'Huyvetter M, Vincke C, Xavier C, Aerts A, Impens N, Baatout S, De Raeve H, Muyldermans S, Caveliers V, Devoogdt N, Lahoutte T. Targeted radionuclide therapy with A 177Lu-labeled anti-HER2 nanobody. Theranostics. 2014 Apr 25;4(7):708-20. doi: 10.7150/thno.8156. eCollection 2014. PMID 24883121
- [Background] Pruszynski M, D'Huyvetter M, Bruchertseifer F, Morgenstern A, Lahoutte T. Evaluation of an Anti-HER2 Nanobody Labeled with 225Ac for Targeted alpha-Particle Therapy of Cancer. Mol Pharm. 2018 Apr 2;15(4):1457-1466. doi: 10.1021/acs.molpharmaceut.7b00985. Epub 2018 Mar 7. PMID 29502411
- [Background] Puttemans J, Dekempeneer Y, Eersels JL, Hanssens H, Debie P, Keyaerts M, Windhorst AD, van der Aa F, Lecocq Q, Breckpot K, Morgenstern A, Bruchertseifer F, Lahoutte T, Devoogdt N, D'Huyvetter M. Preclinical Targeted alpha- and beta--Radionuclide Therapy in HER2-Positive Brain Metastasis Using Camelid Single-Domain Antibodies. Cancers (Basel). 2020 Apr 21;12(4):1017. doi: 10.3390/cancers12041017. PMID 32326199
- [Derived] Zhao L, Liu C, Xing Y, He J, O'Doherty J, Huang W, Zhao J. Development of a 99mTc-Labeled Single-Domain Antibody for SPECT/CT Assessment of HER2 Expression in Breast Cancer. Mol Pharm. 2021 Sep 6;18(9):3616-3622. doi: 10.1021/acs.molpharmaceut.1c00569. Epub 2021 Jul 30. PMID 34328338